CLINICAL TRIAL: NCT06664697
Title: Post-Market Clinical Investigation of the IotaSOFT Insertion System for Use with Cochlear Implant Surgery
Brief Title: Post-Market Clinical Investigation of the IotaSOFT Insertion System
Acronym: ACE
Status: Recruiting | Type: Observational
Sponsor: iotaMotion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICI2401
Record Dates: First submitted 2024-10-07; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss, Cochlear; Cochlear Implantation; Hearing Loss, Sensorineural
Keywords: cochlear implantation; sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Retrospective: Retrospective Review of patient records
  Interventions: Device: Cochlear Implantation with Robotic-Assisted Insertion System
- Prospective: Prospective data collection of subjects receiving a cochlear implant with robotic-assisted cochlear implant
  Interventions: Device: Cochlear Implantation with Robotic-Assisted Insertion System

INTERVENTIONS:
Device: Cochlear Implantation with Robotic-Assisted Insertion System — The purpose of the study is to collect additional safety data in retrospective and prospective subjects who receive a cochlear implant using the iotaSOFT Insertion System.

SUMMARY:
The purpose of the proposed study is to evaluate the continued safety of the iotaSOFT Insertion System when used by a surgeon to assist with inserting a CI electrode array in one ear per subject

DETAILED DESCRIPTION:
available iotaSOFT Insertion System when used per intended use for insertion of a cochlear implant electrode array in subjects 12 years and older. The purpose of the study is to collect additional safety data in retrospective and prospective subjects. The primary object of the study is to demonstrate post-market safe use of the commercially available iotaSOFT Insertion System. The secondary objective of the study is to define procedural characteristics including device deficiencies, electrode array insertion speed, rate of tip fold-over, and objective measures of cochlear implant functionality to demonstrate effective use of the commercially available iotaSOFT Insertion System.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates with sensorineural hearing loss who received or will receive unilateral or bilateral cochlear implantation according to indications for use with FDA approved cochlear implant devices, as listed below:

   1. Advanced Bionics HiFocus SlimJ
   2. Cochlear Slim Straight
   3. MED-EL Flex 24 and 28
2. Age 12 years or older at the time of CI surgery.
3. Willingness to participate in the study and able to comply with the follow-up visit requirements.

Exclusion Criteria:

1. Prior cochlear implantation in the ear to be implanted.
2. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array or present an increased risk of aberrant insertion.
3. Craniofacial abnormality, temporal squamosal skull thickness less than 3mm, major cochlear lesions (e.g., fibrosis, fracture, or ossification), or cochlear malformations.
4. Deafness due to lesions of the acoustic nerve or central auditory pathway.
5. Diagnosis of auditory neuropathy.
6. Active middle-ear infection or tympanic membrane perforation in the presence of active middle ear disease.
7. Absence of cochlear development.
8. Additional medical concerns that would prevent participation in evaluations as determined by the investigator.
9. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the procedure and investigational device.
10. Non-native English speakers who are unable to read, understand and/or speak English for completion of required procedures
11. Planned or current participation in a clinical study of an investigational device or drug.
12. Must not fit the definition of a vulnerable subjects, as per FDA regulations 21 CFR Parts 50 and 56

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A minimum of 50 subjects with sensorineural hearing loss and who have received a cochlear implant using the commercially available iotaSOFT insertion system or are scheduled for unilateral or bilateral cochlear implant surgery will be enrolled, such that a minimum of 50 subjects/ears using iotaSOFT will be attempted
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Experiencing a Serious or Related Adverse Event Due to Use of the iotaSOFT Insertion System During Cochlear Implant Surgery | 1 month post-activation
  Number of Subjects Experiencing a Serious or Related Adverse Event Due to Use of the iotaSOFT Insertion System During Cochlear Implant Surgery through 1 month post-operative follow-up

SECONDARY OUTCOMES:
Number of device deficiencies related to the use of the iotaSOFT Insertion System | 1 month post-activation
  Number of reported device deficiencies related to the use of the iotaSOFT Insertion System at the time of cochlear implant surgery

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Oregon Health and Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Cohort data will be provided for analysis for publication and presentation and individual data points will be pulled for reporting requirements only. Primary and secondary endpoint data will be exported and analyzed for required reporting.
Supporting Information: Study Protocol, SAP, CSR